CLINICAL TRIAL: NCT01964118
Title: Can Intermittent Fasting Mimic the Metabolic and Cardiovascular and Anti-aging Effects of Calorie Restriction?
Acronym: IF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201303081
Record Dates: First submitted 2013-10-07; First posted 2013-10-17 (Estimated); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Obesity; Overweight
Keywords: intermittent fasting; obesity; calorie restriction
MeSH Terms: conditions — Obesity; Overweight; Intermittent Fasting | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Other): The participants randomized to the crossover group begin study participation as a control group (no changes in food intake) for the first 6 months and switch to IF for the remaining 6 months of the study.
  Interventions: Other: control group
- Intermittent Fasting group (Experimental): Participant with a BMI between 28 and 35 kg/m2 will fast 3 non-consecutive days per week, whereas participant with a BMI between 24 and 27.9 kg/m2 will fast 2 non-consecutive days per week. Individuals following intermittent fasting (IF) will work with the study dietitian to design their weekly meal plans and menus for the non-fasting days. The subjects following IF will be asked to skip breakfast, lunch, dinner, snacks, and calorie-containing beverages on the fast days, but we will give them the option to consume at dinner a big salad (i.e. non-starchy raw and/or cooked vegetables dressed with 2 tablespoons of salad dressing prepared with vegetable oil, vinegar and seasonings).
  Interventions: Other: Intermittent Fasting group

INTERVENTIONS:
Other: Intermittent Fasting group — Intermittent fasting for 12 months
  Arms: Intermittent Fasting group
Other: control group — usual diet for 6 months and intermittent fasting for other 6 months
  Arms: Control group

SUMMARY:
The purpose of Intermittent Fasting study is to investigate whether intermittent fasting could decrease the chronic inflammation levels in overweight/obese people.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether or not IF reduces the level of chronic inflammation as evidenced by a decrease in high sensitive C-reactive protein (hsCRP), as the main outcome measure

ELIGIBILITY:
Inclusion Criteria:

* The participants in this study will be 50 men and women in the 30 to 65 year age range, who have a BMI in the high normal to moderately obese range (i.e. 24 to 35 kg/m2),
* Participants who are eating usual US diets and are sedentary to moderately active (i.e. not exercise trained).

Exclusion Criteria:

* History of any chronic disease process that could interfere with interpretation of results
* Smoking, pregnancy, alcoholism, psychiatric problems, life situations that would interfere with study participation and compliance.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in HSCRP ( high sensitivity C-reactive protein) at 6 and 12 months | Every 6 months- baseline, 6 month and 12 month
  HSCRP would be measured in mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Tosti, MD, Principal Investigator — Washington University School of Medicine; Luigi Fontana, MD, Phd, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Only to publish

REFERENCES:
- [Background] Goodrick CL, Ingram DK, Reynolds MA, Freeman JR, Cider NL. Effects of intermittent feeding upon growth and life span in rats. Gerontology. 1982;28(4):233-41. doi: 10.1159/000212538. PMID 7117847
- [Derived] Barve RA, Veronese N, Bertozzi B, Tosti V, Cagigas ML, Spelta F, Cava E, Piccio L, Early DS, Head RD, Fontana L. Cardiometabolic and molecular adaptations to 6-month intermittent fasting in middle-aged men and women with overweight: secondary outcomes of a randomized controlled trial. Nat Commun. 2025 Dec 13;16(1):11370. doi: 10.1038/s41467-025-66366-8. PMID 41390492
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717